CLINICAL TRIAL: NCT05256615
Title: Optimizing Blood Glucose Control in Pregnant Women Diagnosed With Gestational and Type 2 Diabetes Mellitus.
Brief Title: Exercise Timing and Gestational Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00097525
Record Dates: First submitted 2021-12-23; First posted 2022-02-25 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Pregnancy Related; Diabetes; Diabete Mellitus; Type 2 Diabetes; Pre-diabetes; Exercise
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2; Glucose Intolerance; Motor Activity

STUDY DESIGN:
Intervention Model Description: This study comprises of two groups; a diabetes and a non-diabetes group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diabetes (Experimental): Participants recruited to this arm have been clinically diagnosed with either gestational, pre- or type 2 diabetes.
  Interventions: Behavioral: 30-minute walking intervention; Behavioral: 10-minute
- Non-diabetes (Experimental): Participants recruited to this arm of the study do not have gestational, pre- or type 2 diabetes.
  Interventions: Behavioral: 30-minute walking intervention; Behavioral: 10-minute

INTERVENTIONS:
Behavioral: 30-minute walking intervention — Participants are asked to go for a 30 minute walk once per day at any time except the 1 hour after a meal. During these walks they are asked to record heart rate using a heart rate monitor and a phone application.
  Other Names: LONG
Behavioral: 10-minute — Participants are asked to go for a 10-minute walk after each meal occurring 3 times daily. During these walks they are asked to record heart rate using a heart rate monitor and a phone application.

SUMMARY:
The aim of this study is to understand if the timing of exercise around food intake can help improve blood sugar management in pregnant individuals with diabetes.

DETAILED DESCRIPTION:
Between 3 - 20% of women develop gestational diabetes mellitus (GDM) during pregnancy, a condition in which blood sugar control is poor and can have serious health effects for both mom and baby. Women with GDM are at elevated risk of developing dangerously high blood pressure during pregnancy and type 2 diabetes later in life. GDM also puts the baby at an increased risk of excessive birth weight, low blood sugar at birth, and future risk of type 2 diabetes.

The 2019 Canadian Guideline for Physical Activity throughout Pregnancy recommends that women be physically active for at least 150 minutes spread over at least 3 days each week. Managing high blood sugars with exercise improves outcomes for mom and baby; however, optimal timing of exercise has not been investigated.

The goal of this study is to determine if exercising after meals in shorter bouts is more effective at controlling post-meal blood sugars than exercising in larger amounts between meals.

This is a fully remote study; participants will receive all necessary equipment in the mail and all interactions with the researcher will be done via phone, video call and email.

The study will recruit 30 pregnant women diagnosed (or not) with diabetes (gestational, pre-, or type 2 diabetes mellitus) after 20 weeks' gestation to participate in this 2-week study. Following a 2 day baseline period, they will be randomly assigned to: 1) walk for 10 minutes after each meal (SHORT), or 2) walk for 30 minutes once per day at any time except in the hour after eating (LONG) for 5 days. Following a 2- day washout period, women will then complete the alternative exercise protocol for an additional 5 days. Women will wear a Continuous Glucose Monitor to track blood sugars, and an accelerometer to track activity patterns (e.g., compliance to the intervention) for seven consecutive days. The Investigators hypothesize that women who walk for 10 minutes after each meal will have a blunted rise in blood sugar following food intake, compared to the women in the 30- minute walking group. Findings from this novel study may help better treat GDM, improving lifelong health for moms and babies around the world.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age
* singleton pregnancies
* healthy pregnant individuals or diagnosed with gestational, pre- or Type 2 diabetes

Exclusion Criteria:

* less than 18 years of age
* presents with contraindications to prenatal exercise (e.g., preeclampsia)
* multiple pregnancies (i.e. twins, triplets etc.)
* currently taking Metformin

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Due to the topic of this study, this study targets female gender.
Enrollment: 41 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-06-07 (Actual); Study Completion 2024-06-07 (Actual)

PRIMARY OUTCOMES:
Postprandial blood glucose (mmol/l) | Day 1 to Day 14
  Mean, peak and nadir 24 hour daily glucose, glycemic variability, fasting glucose, time spent in hyperglycemia (>10mmol/l), and time spent in hypoglycemia (<3.5mmol/l). These values will be compared between pregnant individuals diagnosed with gestational, pre- or Type 2 diabetes, and healthy pregnant individuals. High postprandial glucose level indicates poor blood glucose control.
Daily physical activity (minutes per day) | Day 1 to Day 14
  All participants will be asked to wear an accelerometer (Actigraph wGT3X-BT Monitor, Actigraph LLC) for fourteen consecutive days to record 24-hour physical activity (min/d). This information will be collected to determine overall physical activity and movement behaviours (including light, moderate and vigorous activity intensity).
Sleep (minutes per night) | Day 1 to Day 14
  All participants will be asked to wear an accelerometer (Actigraph wGT3X-BT Monitor, Actigraph LLC) for fourteen consecutive nights to record 24-hour physical activity (min/d). This information will be collected to determine total sleep time (min/day)

SECONDARY OUTCOMES:
Heart rate (bpm) | Day 3-7 and day 9-14
  Participants will be lent a heart rate monitor chest strap and watch (Polar) to wear during their walking sessions to confirm they are in the prescribed intensity range. The chest strap is worn around the chest with the sensor placed just inferior to the sternum. It wirelessly connects to the watch which displays their heart rate in beats per minute (BPM). Participants are asked to maintain a heart rate 0f 101 - 146 bpm to represent moderate intensity physical activity.
Health history questionnaires | Pre-intervention
  Health history (personal and familial) may affect the results of variables assessed within this study. Participants will be asked about their age (years), height (cm) and weight) (kg). They will also be asked about their pregnancy health and any complications that should be noted. The over all purpose of this questionnaire is to allow us describe the type of participant recruited to this study. This questionnaire can be submitted online via Redcap, or by hard copy (if requested).
Physical activity questionnaires | Pre-intervention
  We will use a questionnaire prior to the intervention to estimate participants physical activity level using the Pregnancy Physical Activity Questionnaire. Total activity time will be computed (min/day) from this. This questionnaire can be submitted online via Redcap, or by hard copy (if requested).
Sleep quality questionnaire | Pre-intervention
  We will use a questionnaire prior to the intervention to estimate participants sleep quality using the Pittsburgh Sleep Quality Index. This questionnaire can be submitted online via Redcap, or by hard copy (if requested). Each component is scored on a scale of 0-3 with higher values representing greater sleep dysfunction.
Food Diary | Days 1 - 14
  Diet may affect the results of variables assessed within this study. We will ask participants to keep a hand written diary log for the duration of the study about the type and amount (grams) of food intake they are consuming.
Maternal outcomes | Through study completion - an average of 1 year postpartum
  Data on maternal complications if any, will be recorded from medical notes. This may include although not limited to diagnosis of pre-eclampsia, hypertension in pregnancy, caesarean section, birth complications, instrumental delivery, blood loss, and length of labour. These outcomes will be collected as categorical variables with 'yes ' or 'no' as an answer.
Infant outcomes | Through study completion - an average of 1 year postpartum
  Data on infant outcomes will be recorded from medical notes. This may include although not limited to weeks of gestation at birth, birth weight, hypoglycemia at birth, admission to NICU, breastfeeding status, infant mortality, and 2-month development. These outcomes will be collected as categorical variables with 'yes ' or 'no' as an answer.
Infant Apgar Scores | Through study completion - an average of 1 year postpartum
  Apgar scores will be collected from medical notes. An apgar score

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No